CLINICAL TRIAL: NCT01161498
Title: A Phase 3 Randomized Trial of Concurrent Cisplatin & Radiotherapy With Or Without ONCOVEX^GM-CSF In Previously Untreated Patients With Locally Advanced Squamous Cell Carcinoma Of The Head And Neck
Brief Title: Study of Safety and Efficacy of Talimogene Laherparepvec With Cisplatin and Radiotherapy for Treatment of Locally Advanced Head and Neck Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The changing aetiology of squamous cell carcinoma of the head and neck (SCCHN).
Sponsor: BioVex Limited (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 006/09; 20110130 (Other: Amgen Inc.)
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Squamous Cell Carcinoma; Head and Neck Cancer
Keywords: squamous cell; OncoVEX^GM-CSF; Oncovex; chemoradiation; Cisplatin
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms | interventions — talimogene laherparepvec; Radiation; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation/Cisplatin (Active Comparator): Participants received cisplatin (100 mg/m²) administered intravenously on Days 0, 21, and 42. Radiation was administered concurrently with cisplatin in 35 fractions over a 7-week period.
  Interventions: Radiation: Radiation; Drug: Cisplatin
- Talimogene Laherparepvec + Radiation/Cisplatin (Experimental): The first dose of talimogene laherparepvec was up to 8 mL total volume (up to 4 mL per lesion) at 10⁶ plaque-forming units (PFU)/mL, administered into all injectable affected nodes on Day 0. Subsequent doses were up to 8 mL total volume (up to 4 mL per lesion) at 10⁸ PFU/mL on Days 21, 42, and 63. Participants also received cisplatin (100 mg/m²) administered intravenously on Days 0, 21, and 42 and radiation administered concurrently in 35 fractions over a 7-week period.
  Interventions: Biological: Talimogene Laherparepvec; Radiation: Radiation; Drug: Cisplatin

INTERVENTIONS:
Biological: Talimogene Laherparepvec — Administered by intratumoral injection
  Other Names: OncoVEX^GM-CSF; IMLYGIC
  Arms: Talimogene Laherparepvec + Radiation/Cisplatin
Radiation: Radiation — 70 grays of radiation administered in 35 fractions over 7 weeks
Drug: Cisplatin — Administered by intravenous infusion

SUMMARY:
This study is being conducted to learn about the safety and risks of using talimogene laherparepvec to treat patients with head and neck cancer and to see if talimogene laherparepvec and chemoradiation together can destroy the tumours versus the use of chemoradiation alone. This study may provide information on the usefulness of talimogene laherparepvec combined with chemoradiation as a future treatment for head and neck cancer.

DETAILED DESCRIPTION:
The objective is to evaluate the efficacy and safety of treatment with chemoradiation (CRT) plus talimogene laherparepvec compared to CRT alone in previously untreated patients with locally advanced squamous cell carcinoma of the head and neck (SCCHN) for which surgical resection is not clinical indicated. The efficacy endpoints of the study aim to demonstrate overall clinical benefit for patients treated with talimogene laherparepvec as compared to CRT alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years
2. Eastern Co-Operative Oncology Group (ECOG) Performance Status ≤ 1
3. Histological evidence (from the primary lesion and/or lymph nodes) of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx
4. Stage III or IV disease (T2N2-3M0, T3-4N1-3M0)
5. No evidence of distant metastases by computed tomography (CT) or positron emission tomography (PET)/CT scan
6. Life expectancy > 4 months
7. Neutrophil count ≥ 2,000/mm^3
8. Platelet count ≥ 100,000/mm^3
9. Hemoglobin ≥ 10 g/dL
10. Bilirubin ≤ 1.5 times upper limit of normal (ULN)
11. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN
12. Alkaline phosphatase ≤ 2.5 times ULN
13. Creatinine clearance ≥ 60 mL/min
14. Female patients of child-bearing potential (i.e. not surgically sterile, or not having spontaneous amenorrhea for at least 12 months) must agree to use an effective form of contraception during the treatment phase of the study.
15. Male patients must agree to use a condom with spermicide or their female partner must use an effective method of birth control.
16. Provide written informed consent in accordance with all applicable regulations and follow the study procedures. Patients must be capable of understanding the investigational nature, potential risks and benefits of the study.

Exclusion Criteria:

1. Prior treatment for locally advanced SCCHN (No prior surgery for SCCHN except nodal sampling or biopsy for study disease).
2. Patients with T1-2N1 or T1N2-3.
3. Pre-existing peripheral neuropathy ≥ Grade 2 (motor or sensory).
4. Weight loss > 20% of body weight within 3 months of screening (unless purposeful).
5. Surgery ≤ 28 days before randomization with the exception of feeding tube placement, dental extractions, central venous catheter placement, biopsies and nodal sampling.
6. Cancer of the nasopharynx, sinus, salivary gland or skin.
7. Previous radical radiation therapy (RT) to the head and neck region, excluding superficial RT for a non-melanomatous skin cancer.
8. Prior cancers, except: those diagnosed > 5 years ago with no evidence of disease recurrence and clinical expectation of recurrence of less than 5%; or successfully treated non-melanoma skin cancer; or carcinoma in situ of the cervix.
9. Significant intercurrent illness that will interfere with the chemotherapy or radiation therapy such as human immunodeficiency (HIV) infection, cardiac failure, pulmonary compromise (chronic obstructive pulmonary disease, pneumonia or respiratory decompensation) resulting in hospitalization within 12 months of screening, or active infection.
10. Any significant cardiac disease (e.g., New York Heart Association (NYHA) Class 3 or 4; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty or coronary artery bypass graft (CABG) within the past 6 months; or uncontrolled atrial or ventricular cardiac arrhythmias..
11. High risk for poor compliance with therapy or follow up as assessed by the investigator.
12. Active herpes labialis, other lesions due to herpes simplex virus type I (HSV1) or dermatoses involving or within 50 cm of the lesions to be injected; active HSV1 lesions must have resolved before talimogene laherparepvec is injected.
13. Prior systemic chemotherapy for any type of cancer.
14. Patients for whom radiation therapy is contraindicated.
15. Pregnant or breast-feeding female. Confirmation that women of child-bearing potential are not pregnant. A negative serum β- human chorionic gonadotropin (β-hCG) pregnancy test result must be obtained during the screening period.
16. Currently enrolled and receiving an investigational agent in a clinical research study or received an investigational agent for any reason within 4 weeks prior to screening.
17. Require intermittent or chronic treatment with an anti-herpetic drug (e.g., acyclovir), other than intermittent topical use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Harrington, MD, Principal Investigator — Royal Marsden, UK
Locations (6):
- United States (5):
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - James Graham Brown Cancer Center, University of Louisville, Louisville, Kentucky
  - Gabrail Cancer Center, Canton, Ohio
  - Medical Univesity of South Carolina, Charleston, South Carolina
  - VCU Massey Cancer Center, Richmond, Virginia
- The Royal Marsden Hospital, London, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to patients with advanced, non-metastatic, stage III or IV squamous cell carcinoma of the head and neck (SCCHN).
Period: Overall Study
Arm/Group | Radiation/Cisplatin | Talimogene Laherparepvec + Radiation/Cisplatin
Started | 3 | 2
Completed | 3 | 1
Not Completed | 0 | 1
Not completed — Disease Progression | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Talimogene Laherparepvec + Radiation/Cisplatin: The first dose of talimogene laherparepvec was up to 8 mL total volume (up to 4 mL per lesion) at 10⁶ PFU/mL, administered into all injectable affected nodes on Day 0. Subsequent doses were up to 8 mL total volume (up to 4 mL per lesion) at 10⁸ PFU/mL on Days 21, 42, and 63. Participants also received cisplatin (100 mg/m²) administered intravenously on Days 0, 21, and 42 and radiation administered concurrently in 35 fractions over a 7-week period.
- Total: Total of all reporting groups
Arm/Group | Radiation/Cisplatin | Talimogene Laherparepvec + Radiation/Cisplatin | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: 2-year Event-free Survival
Description: Event-free survival is defined as the time from randomization until the first evidence of relapse, disease progression (local, regional, metastatic, or second primary), or death from any cause. Because this study was terminated with only 5 participants enrolled, and the study was terminated in the first year, this endpoint was not analyzed.
Time Frame: 2 years
Arm/Group | Radiation/Cisplatin | Talimogene Laherparepvec + Radiation/Cisplatin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Clinical Objective Response (cOR)
Description: Tumor response was assessed by computed tomography (CT) scan according to a modified version of the revised Response Evaluation Criteria In Solid Tumors (RECIST) criteria (version 1.1). Objective response is defined as achieving a clinical partial response (cPR) or complete response (cCR). cCR is defined as disappearance of all baseline lesions. Any pathological lymph nodes must have a reduction in short axis to < 10 mm. cPR is defined as at least a 30% decrease in the sum of diameters of baseline lesions. Progressive disease (PD) is defined as at least a 20% increase in the sum of diameters of baseline lesions, taking as reference the smallest sum on study, and an absolute increase of at least 5 mm, or the appearance of any new lesions.
  Because this study was terminated with 5 patients enrolled, data for this endpoint were summarized in by-patient listings only and the cOR rate was not calculated. Therefore a summary of response at the end of study is reported.
Time Frame: End of trial; the maximum time on study was 20 weeks.
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Radiation/Cisplatin | Talimogene Laherparepvec + Radiation/Cisplatin
Number analyzed (Participants) | 3 | 2
participants
  Clinical Complete Response (cCR) | 2 | 1
  Clinical Partial Response (cPR) | 0 | 0
  Progressive Disease | 1 | 0
  Unevaluable | 0 | 1

3. Secondary Outcome: Metabolic Complete Response (mCR)
Description: Response to therapy was assessed using [(18)F] fluorodeoxyglucose positron emission tomography (FDG PET) imaging to detect metabolically active tumors.
  Metabolic complete response (mCR) is defined as complete disappearance of FDG uptake attributable to tumor compared to baseline scan.
  Partial metabolic response (mPR) is defined as a > 40% decrease in specific uptake compared to the initial value in over half of the lesions.
  Disease progression (mPD) is defined as a specific uptake increase in any lesion, appearance of new lesions, or presence of extended areas of disease activity.
  Stable metabolic response (mSD) is defined as a decrease in uptake < 40% of the initial value of over half the lesions.
  Because this study was terminated with 5 patients enrolled, data for this endpoint were summarized in by-patient listings only and the metabolic complete response rate was not calculated. Therefore a summary of metabolic response at end of study is reported.
Time Frame: End of study; the maximum time on study was 20 weeks.
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Radiation/Cisplatin | Talimogene Laherparepvec + Radiation/Cisplatin
Number analyzed (Participants) | 3 | 2
participants
  Metabolic Complete Response (mCR) | 1 | 1
  Metabolic Partial Response (mPR) | 0 | 0
  Metabolic Progressive Disease (mPD) | 1 | 0
  Stable Metabolic Response (mSD) | 0 | 0
  Unevaluable | 1 | 1

4. Secondary Outcome: Pathologic Complete Response (mCR)
Description: Response to therapy was assessed histopathologically from biopsies taken at surgery for those participants who had surgery prior to Week 22.
  If no viable tumor cells were identified in surgical specimens (where the patient had surgery) the patient was classified as having a pathological complete response (pCR), and if viable tumor cells were identified, the patient was classified as having an incomplete pathologic response.
  Because this study was terminated with 5 patients enrolled, data for this endpoint were summarized in by-patient listings only and the pathologic complete response rate was not calculated. Therefore a summary of participants with a pathologic complete response before the end of study is reported.
Time Frame: Up to Week 20
Population: Randomized participants who had protocol-specified surgery
Measure: Number; unit: participants
Arm/Group | Radiation/Cisplatin | Talimogene Laherparepvec + Radiation/Cisplatin
Number analyzed (Participants) | 1 | 0
participants | 0 |

5. Secondary Outcome: Time to Locoregional Failure
Description: Locoregional failure is defined as disease progression in the head and neck area at any time following completion of chemoradiotherapy.
  Because this study was terminated with 5 subjects enrolled, time to locoregional failure was not analyzed.
Time Frame: Up to 27 months
Arm/Group | Radiation/Cisplatin | Talimogene Laherparepvec + Radiation/Cisplatin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Distant Failure
Description: Distant failure is defined as disease progression at any site other than the head and neck area at any time following completion of chemoradiotherapy.
  Because this study was terminated with 5 participants enrolled, time to distant failure was not analyzed.
Time Frame: Up to 27 months
Arm/Group | Radiation/Cisplatin | Talimogene Laherparepvec + Radiation/Cisplatin
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to Any Failure
Description: Any failure is defined as disease progression at any site at any time following completion of chemoradiotherapy.
  Because this study was terminated with 5 participants enrolled, time to any failure was not analyzed.
Time Frame: Up to 27 months
Arm/Group | Radiation/Cisplatin | Talimogene Laherparepvec + Radiation/Cisplatin
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death from any cause.
  Because this study was terminated with 5 participants enrolled, overall survival was not analyzed.
Time Frame: Up to 5 years after chemoradiotherapy
Arm/Group | Radiation/Cisplatin | Talimogene Laherparepvec + Radiation/Cisplatin
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Disease-specific Survival
Description: Disease-specific survival is defined as the time from randomization to death of the patient due to the cancer under study.
  Because this study was terminated with 5 participants enrolled, disease-specific survival was not analyzed.
Time Frame: Up to 5 years after chemoradiotherapy
Arm/Group | Radiation/Cisplatin | Talimogene Laherparepvec + Radiation/Cisplatin
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Participants With N1-2 Disease at Baseline Requiring Neck Dissection
Description: Participants with Baseline Nl or N2 disease (lymph node metastasis not more than 6 cm in greatest dimension) with persistent disease as determined at the post chemoradiotherapy assessment of response were to proceed to neck dissection as permitted by the institution no later than Week 22. Since this study terminated prematurely neck dissection data were not collected or analyzed.
Time Frame: Weeks 19 - 21
Arm/Group | Radiation/Cisplatin | Talimogene Laherparepvec + Radiation/Cisplatin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Radiation/Cisplatin | Talimogene Laherparepvec + Radiation/Cisplatin
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation/Cisplatin (N=3) | Talimogene Laherparepvec + Radiation/Cisplatin (N=2)
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation/Cisplatin (N=3) | Talimogene Laherparepvec + Radiation/Cisplatin (N=2)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1
Saliva altered (Gastrointestinal disorders) | 1 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Catheter site erythema (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.